CLINICAL TRIAL: NCT06758778
Title: An Open-Label, Balanced, Randomized, Single Dose, Two-Treatment, Two-Sequence, Two-Period ,Two-Way Crossover Oral Bioavailability Study of CreNeuroSTM CNS Fish Oil Plus Softgels [Eicosapentaenoic Acid (as Ethyl Ester) 342 mg; L-5-methyltetrahydrofolate 1.875 mg; Other Vitamins and Minerals] (Test Product) Compared With Co-administration of Icosapent Ethyl 1000 mg Capsules (Reference Product-1) and L-methylfolate Calcium 7.5 mg Capsules (Reference Product-2) in Healthy Human Adult Subjects Under Fasting Conditions
Brief Title: CreNeuroS™️CNS Fish Oil Plus Softgels Compared to Vascepa® Capsules and Deplin® Capsules in a Pharmacokinetic, Single Dose Evaluation on Healthy Adult Human Subjects Under Fasting Conditions
Acronym: BE-001-2024
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Credit Pharmaceutical Co., Ltd. (Industry)
Collaborators: Glogen Clinical Research Pvt. Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BE-001-2024
Record Dates: First submitted 2024-12-23; First posted 2025-01-06 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Bioavailability
MeSH Terms: interventions — Minerals; eicosapentaenoic acid ethyl ester; Capsules; 5-methyltetrahydrofolate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CreNeuroS CNS Fish Oil Plus Softgel (Experimental): CreNeuroS CNS Fish Oil Plus Softgel [380 mg of fish oil contains Eicosapentaenoic Acid (EPA) （as EE）342 mg; L-5- Methyltetrahydrofolate 1.875 mg; other Vitamins and Minerals] Distributed by: Fidelity Biopharma Co., USA.
  Interventions: Dietary Supplement: CreNeuroS CNS Fish Oil Plus Softgel [380 mg of fish oil contains Eicosapentaenoic Acid (EPA) （as EE）342 mg; L-5- Methyltetrahydrofolate 1.875 mg; other Vitamins and Minerals]
- Reference Product (Active Comparator): Reference product (R1): Vascepa® (Icosapent ethyl) 1000 mg Capsules Manufactured by：Patheon Softgels B.V. Reference product (R2): Deplin® (L-methylfolate Calcium) 7.5 mg Capsules Manufactured by：Alfasigma USA, Inc.
  Interventions: Dietary Supplement: Vascepa® (Icosapent ethyl) 1000 mg Capsules, Deplin® (L-methylfolate Calcium) 7.5 mg Capsules

INTERVENTIONS:
Dietary Supplement: CreNeuroS CNS Fish Oil Plus Softgel [380 mg of fish oil contains Eicosapentaenoic Acid (EPA) （as EE）342 mg; L-5- Methyltetrahydrofolate 1.875 mg; other Vitamins and Minerals] — Test product
  Arms: CreNeuroS CNS Fish Oil Plus Softgel
Dietary Supplement: Vascepa® (Icosapent ethyl) 1000 mg Capsules, Deplin® (L-methylfolate Calcium) 7.5 mg Capsules — Reference product
  Arms: Reference Product

SUMMARY:
The objective of this study is to evaluate the oral bioavailability of 'CreNeuroS CNS Fish Oil Plus Softgels [Eicosapentaenoic Acid (as Ethyl Ester) 342 mg; L-5-methyltetrahydrofolate 1.875 mg; other Vitamins and Minerals] (Test Product) compared with co-administration of Omega-3-acid Ethyl ester 1000 mg Capsules (Reference Product-1) and L-methylfolate Calcium 7.5 mg Capsules (Reference Product-2) in healthy human adult subjects under fasting conditions.

DETAILED DESCRIPTION:
This is an Open-Label, Balanced, Randomized, Single Dose, Two-Treatment, Two-Sequence, Two-Period ,Two-Way Crossover oral Bioavailability study of CreNeuroSTM CNS Fish Oil Plus Softgels [Eicosapentaenoic Acid (as Ethyl Ester) 342 mg; L-5-methyltetrahydrofolate 1.875 mg; other Vitamins and Minerals] (Test Product) compared with co-administration of Omega-3-acid Ethyl ester 1000 mg Capsules (Reference Product-1) and L-methylfolate Calcium 7.5 mg Capsules (Reference Product-2) in healthy human adult subjects under fasting conditions.

A total number of 14 normal healthy adult human subjects will be included in the study.

A total of 35 blood samples will be collected from each subject in each study period.

There will be atleast 28 days washout period between two treatments in the study.

The following analytes will be determined in plasma using a validated LC-MS/MS (Liquid chromatography tandem mass spectrometry) method.

* Total Eicosapentaenoic Acid (EPA) in plasma
* L-5-methyltetrahydrofolate (L-5-MTHF) in plasma

ELIGIBILITY:
Inclusion Criteria:

* • Healthy human subjects aged between 18 and 45 years (including both).

  * Subjects with a BMI between 18.50-25.00 Kg/m2 (including both) but body weight not less than 50 Kgs.
  * Subjects with normal health as determined by personal medical history, Clinical examination and laboratory examinations including serological tests during the screening as per section 5.3.
  * Subjects having normal 12-lead electrocardiogram (ECG).
  * Subjects having normal chest X-Ray (P/A view) whose X-Ray was taken not more than 180 days prior to the check-in of Period-I.
  * Subjects able to communicate effectively.
  * Subjects willing to give written informed consent and adhere to all the requirements of this protocol.
  * Subject is a non-smoker or moderate smoker (not more than 10 cigarettes or beedis/day).
  * Subject is a non-alcoholic or non-alcoholic abuse (Alcohol abuse will be defined as >14 drinks per week (1 drink=360 mL beer, 150 mL wine or 45 mL hard liquor).
  * Additional inclusion criteria for female subjects, Female of childbearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD) or abstinence: or Surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy has been performed on the subject).

Exclusion Criteria:

* • Subjects having contraindications or hypersensitivity to study drug or related group of drugs.

  * An unusual or abnormal diet, for whatever reason within 48.00 hours prior to admission of each period, e.g., fasting due to religious reasons.
  * History of Hypertension.
  * History of dehydration from diarrhea, vomiting or any other reason within a period of 24.00 hours prior to study admission of each study period.
  * Positive results for drugs of abuse (benzodiazepines, cocaine, opioids, amphetamines, cannabinoids and barbiturates) in urine during the admission of each study period.
  * Positive results for alcohol consumption during the admission of each study period.
  * Intolerance to venipuncture.
  * History or presence of any medical condition or disease according to the opinion of the physician.
  * History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
  * Difficulty with donating blood.
  * Major illness during 90 days before check-in.
  * Participation in a drug Research study within past 90 days of check-in.
  * Donation of blood (i.e. one unit or 350 mL) in the past 90 days before check-in.
  * Difficulty in swallowing solid dosage forms like tablets or capsules.
  * Additional exclusion criteria for female subjects, Volunteer demonstrating a positive pregnancy test. Volunteers who are pregnant, currently breast-feeding or who are likely to become pregnant during the study.

Volunteers who have used implanted or injected hormonal contraceptives anytime during the 6 months prior to study or used hormonal contraceptives within 14 days before dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Baseline-adjusted total eicosapentaenoic acid and baseline-adjusted L-5-methyltetrahydrofolate | Pharmacokinetic plasma samples collected over 432.00 hours (Eicosapentaenoic acid) and 16 hours (L-5-methyltetrahydrofolate) period
  AUC (Area under curve)

SECONDARY OUTCOMES:
Baseline-adjusted total eicosapentaenoic acid and baseline-adjusted L-5-methyltetrahydrofolate | Pharmacokinetic plasma samples collected over 432.00 hours (Eicosapentaenoic acid) and 16 hours (L-5-methyltetrahydrofolate) period
  Tmax (Time to achieve maximum plasma concentration)

CONTACTS AND LOCATIONS:
Locations (1):
- GloGen Clinical Research Pvt. Ltd., Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rusca A, Di Stefano AF, Doig MV, Scarsi C, Perucca E. Relative bioavailability and pharmacokinetics of two oral formulations of docosahexaenoic acid/eicosapentaenoic acid after multiple-dose administration in healthy volunteers. Eur J Clin Pharmacol. 2009 May;65(5):503-10. doi: 10.1007/s00228-008-0605-4. Epub 2009 Jan 16. PMID 19148629
- See also: Pharmacokinetic study on the utilisation of 5-methyltetrahydrofolate and folic acid in patients with coronary artery disease — https://pmc.ncbi.nlm.nih.gov/articles/PMC1574248/